CLINICAL TRIAL: NCT04172389
Title: Multicentric Retrospective Evaluation of the Vesico-vaginal Fistula Repair by Robot Assisted Laparoscopy
Brief Title: Treatment of Vesico-vaginal Fistula by a Robot Assisted Laparoscopy : Results of a Multicentric Series (FFVLARO)
Acronym: FFVLARO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI229
Record Dates: First submitted 2019-11-16; First posted 2019-11-21 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-10

CONDITIONS: Vesico-vaginal Fistula
MeSH Terms: conditions — Vesicovaginal Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: vesico-vaginal fistula robot assisted laparoscopic repair — realization of O'conor technique or extra-vesical technique for vaginal vesico fistula repair in robot assisted coelioscopy

SUMMARY:
Robot-assisted Vesico-Vaginal fistula (VVF) repair was described a few years ago as an alternative to the open approach to minimize the morbidity of this surgery. Very little series have reported the results of robotic VVF repair. The objective of this work was to evaluate the results of robotic VVF repair.

ELIGIBILITY:
Inclusion Criteria:

* presence of a vesico-vaginal fistula

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent a robotic vesico-vaginal fistula repair
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of urinary leakage through the vagina post surgery after the removal of the urinary tube | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: pierre lecoanet, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- centralHNF, Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: No